CLINICAL TRIAL: NCT02406417
Title: The Use of Reflex Strategies and Reflective Testing in the Clinical Chemistry Laboratory for Early Detection of Pituitary Dysfunction in Patients From Primary Care.
Brief Title: Reflective Testing for Early Diagnosis of Pituitary Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not require ethics Approval as it was not considered research.
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RTFPI2015
Record Dates: First submitted 2015-03-02; First posted 2015-04-02 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2015-03

CONDITIONS: Pituitary Dysfunction
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigation for pituitary dysfunction (Experimental): Further investigation for pituitary dysfunction by blood tests, dynamic function tests and pituitary imaging e.g. CT Scan with contrast. Patients identified as being at high risk of having pituitary dysfunction based on preliminary blood tests will have further tests added. If these results point to a likely pituitary dysfunction, the patient will be referred to the Endocrine team for further investigations including dynamic function tests and/or imaging.
  Interventions: Device: Investigation for pituitary dysfunction by blood tests.; Device: Dynamic function tests and pituitary imaging

INTERVENTIONS:
Device: Investigation for pituitary dysfunction by blood tests. — Blood tests for pituitary function (one or more of the following tests: cortisol, LH, FSH, TSH, FT4, testosterone, prolactin) will be added to samples from patients identified as being at high risk from their initial blood results.
Device: Dynamic function tests and pituitary imaging — Patients identified as being highly likely to have a pituitary dysfunction from the results of the blood tests for pituitary function added, will be referred to the Endocrine team for further tests in the form of dynamic function tests and pituitary imaging.

SUMMARY:
Early detection and management of pituitary dysfunction reduces the morbidity that ensues as a consequence of missed or delayed diagnosis of this condition, and which may result in life-threatening events and increased mortality.

The investigators study will explore the use of reflex strategies within the laboratory in capturing suspicious pituitary function test results from Primary Care patients and following these up with appropriate reflective testing. Subsequently patients identified from these results to have a possible underlying piuitary dysfunction will have an alert sent to their family physician prompting referral to the Endocrine team for further investigation and management.

ELIGIBILITY:
Inclusion Criteria:

* Patients from Primary Care found to have one or more abnormal pituitary function test picked up by the laboratory information system in the Clinical Chemistry laboratory.

Exclusion Criteria:

* Patients with known pituitary dysfunction or on medication that may affect pituitary function tests.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
Number of patients found to have biochemical evidence of possible pituitary dysfunction | One year

SECONDARY OUTCOMES:
Number of patients from primary outcome found to have true pituitary dysfunction | 6- 12 months